CLINICAL TRIAL: NCT07147205
Title: Evaluation of Meaning-centered Group Psychotherapy in Integrative Medicine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-0994; NCI-2025-06343 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-08-27; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Psychotherapy; Integrative Medicine
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention with Meaning-Centered Group Psychotherapy (Experimental)
  Interventions: Other: Therapy

INTERVENTIONS:
Other: Therapy — MCGP will be delivered in 8 weekly sessions for 90 minutes over Zoom by a licensed doctoral level psychologist.

SUMMARY:
To learn more about your experience participating in a virtual Meaning-Centered Psychotherapy group.

DETAILED DESCRIPTION:
Primary Objectives

The objectives are to describe the characteristics and outcomes of participants who attend at least one session of MCGP:

1. Describe demographic, clinical characteristics, reasons for referral, and IMC utilization data for participants who attend MCGP.
2. Examine anxiety, depression, quality of life, meaning in life, and fear of cancer recurrence before and after participation in MCGP.
3. Describe satisfaction and qualitative feedback from group participants, including perceived effectiveness and outcomes, experiences participating in the group virtually, and reactions to specific elements of the therapy modified for cancer survivors, length of group (90 minutes), and the nature of a closed group within the IMC.

   Secondary Objectives
4. Examine whether demographic, clinical, or symptoms-based (pre) measures are associated with number of MCGP sessions attended.
5. Examine whether number of sessions attended is associated with change in outcome measures.

ELIGIBILITY:
Eligibility Criteria

1. Age 18 or older.
2. Male or female.
3. Diagnosis or history of malignant cancer (excluding non-melanoma skin cancer) or tumor disease.
4. Able to read, write, and speak in English.
5. Has access to iOS or Android smartphone, computer, or tablet or device capable of logging onto Zoom.
6. Referred to the Integrative Medicine Clinic, completed consult with IMC physician, referred to health psychology and completed health psychology assessment.
7. Participates in at least one MCGP group session.
8. Willing to review informed consent statement and agree to complete questionnaires.

Exclusion Criteria

1. Children will not be enrolled in this study.
2. Pregnant women will not be enrolled in this study.
3. Cognitively impaired subjects will not be enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Self-report Questionnaires | Through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Conti, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org